CLINICAL TRIAL: NCT00264420
Title: A Phase I Pilot Trial to Study the Safety and Efficacy of Concomitant Radiotherapy and Zoledronic Acid for the Palliation of Bone Metastases From Breast Cancer, Prostate Cancer and Lung Cancer
Brief Title: Safety and Efficacy Study of Concomitant Radiotherapy and Zoledronic Acid for Bone Metastases Palliation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Novartis (Industry)
Responsible Party: Dawn Miller, Program Coordinator, Cleveland Clinic Foundation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB7743; Case 8Y04
Record Dates: First submitted 2005-12-06; First posted 2005-12-12 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Bone Metastases; Breast Cancer; Lung Cancer; Prostate Cancer
Keywords: bone metastases; breast cancer; lung cancer; prostate cancer; zoledronic acid; radiation therapy
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms | interventions — Zoledronic Acid

ARMS (1):
- 1 (Experimental): zoledronic acid plus radiation therapy
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — At baseline 4 mg IV zoledronic acid over 15 min. every 4 weeks for 6 months plus radiation therapy 30 Gy in 10 fractions (5 times per week for first two weeks)

SUMMARY:
Zoledronic acid (Zometa) belongs to a class of drugs called bisphosphonates. Bisphosphonates are used in bone metastases to keep the cancerous lesion under control in the bone and to help prevent calcium level elevations in the blood. Cancer cell-culture studies at the Cleveland Clinic showed that zoledronic acid and radiation together have more cell killing effect than either one used alone. The purpose of this study is to monitor the healing of bone lesions when using zoledronic acid together with radiation treatment.

DETAILED DESCRIPTION:
Bone metastases are frequently one of the first signs of disseminated disease in cancer patients. Skeletal complications due to metastatic disease include (severe) bone pain, impaired mobility, spinal cord compression, pathological fractures, and hypercalcemia. Radiotherapy and surgery are the options for the specific local treatment of bone metastases. Chemotherapy, hormonotherapy and bisphosphonates are systemic weapons used in the treatment of bone metastases with or without hypercalcemia. Cancers with propensity to metastasize to bones such as breast, prostate, lung and myeloma may possess the capacity to interact with osteoclasts. Osteoclasts are specialized bone cells, which erode mineralized bone by secreting acids and lysosomal enzymes. In normal bone remodeling, osteoclastic bone resorption is coupled to and is in equilibrium with osteoblastic bone formation. The lytic bone destruction associated with malignant bone metastases develops because tumor cells synthesize and release soluble factors that stimulate osteoclasts to resorb bone. The malignant activation of osteoclasts results in a disruption of normal bone remodeling wherein the equilibrium between bone resorption and bone formation is shifted toward increased bone resorption. This relative increase in osteoclastic bone resorption results in a net loss of bone.

Zoledronic acid (Zometa®, CGP42446) is a member of a class of compounds known as bisphosphonates. Bisphosphonates are effective inhibitors of osteoclastic bone resorption. They have therapeutic efficacy in the treatments of hypercalcemia of malignancy, lytic bone disease associated with multiple myeloma, and mixed lytic and blastic bone metastases associated with breast cancer, prostate cancer and lung cancer. In the clinical setting, zoledronic acid is the most potent bisphosphonate.

Conventionally, external beam radiotherapy (RT) is a primary treatment method for the palliation of bone metastases. The aim of RT in bone metastases treatment is to eradicate malignant cells without damaging surrounding normal cells. RT is typically given to the lesion area, in order to spare as much bone marrow as possible. RT is indicated in solitary, lytic and painful bone lesions of multiple myeloma as well as bone metastases from solid tumors such as breast, prostate and lung cancer to prevent the fracture risk or to relieve the pain.

The goal of this study will be to evaluate the safety and efficacy of concomitant standard RT and standard zoledronic acid on the bone metastases of breast, prostate or lung cancer patients. We chose zoledronic acid to use in this study, as it is the most effective FDA approved aminobisphosphonate.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* biopsy proven breast, lung, and/or prostate cancer
* boney metastases with an indication for radiation, either diagnosed radiologically or biopsy proven
* Karnofsky Performance Status >60
* Life expectancy of at least 6 months
* Serum creatinine level ≤ 2.0 mg/dL and calculated creatinine clearance of > 60 mL/min
* Leukocyte count ≥ 3500/mm3
* Hemoglobulin > 11 g/dl
* Platelets > 100,000 / mm3
* Total bilirubin < 2.5 mg/dl

Exclusion Criteria:

* pregnant and lactating women (breast and lung cancer)
* hormonotherapy started less than 3 months prior to randomization (prostate cancer)
* history of allergic reactions to bisphosphonates
* receiving concomitant nephrotoxic chemotherapy
* participation in another clinical trial with an investigational drug or completed an investigational drug trial within the past 30 days
* liver function tests > 1.5 times normal values
* IV calcitonin administration less than 30 days prior to randomization
* laboratory evidence of renal disease
* previous RT to the region of bone metastasis which will be treated in this study
* currently receiving oral or IV bisphosphonate therapy
* presence of ascites
* clinically significant electrocardiographic changes
* hypercalcemia, pathologic fracture, or epidural spinal cord compression
* other organ metastasis
* known hypersensitivity to Zometa® (zoledronic acid) or other bisphosphonates
* current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* recent (within 6 weeks) or planned dental or jaw surgery (e.g.. extraction, implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-12; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
PET-CT | baseline and 6 months

SECONDARY OUTCOMES:
X-ray, baseline | 3 months, 6 months
physical exam | Radiaton Oncology - visits 1, 14, 17
physical exam | Medical Oncology - visits 1, 13, 17

CONTACTS AND LOCATIONS:
Overall Officials: Roger Macklis, MD, Principal Investigator — The Cleveland Clinic

REFERENCES:
- [Background] Fulfaro F, Casuccio A, Ticozzi C, Ripamonti C. The role of bisphosphonates in the treatment of painful metastatic bone disease: a review of phase III trials. Pain. 1998 Dec;78(3):157-169. doi: 10.1016/S0304-3959(98)00135-3. PMID 9870569
- [Background] ABRAMS HL, SPIRO R, GOLDSTEIN N. Metastases in carcinoma; analysis of 1000 autopsied cases. Cancer. 1950 Jan;3(1):74-85. doi: 10.1002/1097-0142(1950)3:13.0.co;2-7. No abstract available. PMID 15405683
- [Background] Scher HI, Chung LW. Bone metastases: improving the therapeutic index. Semin Oncol. 1994 Oct;21(5):630-56. No abstract available. PMID 7939753
- [Background] Brown JE, Neville-Webbe H, Coleman RE. The role of bisphosphonates in breast and prostate cancers. Endocr Relat Cancer. 2004 Jun;11(2):207-24. doi: 10.1677/erc.0.0110207. PMID 15163299
- [Background] Lipton A, Berenson JR. Bisphosphonate treatment of lytic bone metastases. Drugs Aging. 1999 Apr;14(4):241-6. doi: 10.2165/00002512-199914040-00001. PMID 10319239
- [Background] Body JJ. Clinical research update: zoledronate. Cancer. 1997 Oct 15;80(8 Suppl):1699-701. doi: 10.1002/(sici)1097-0142(19971015)80:8+3.3.co;2-a. PMID 9362440
- [Background] Mundy GR, Wilkinson R, Heath DA. Comparative study of available medical therapy for hypercalcemia of malignancy. Am J Med. 1983 Mar;74(3):421-32. doi: 10.1016/0002-9343(83)90961-0. PMID 6219578
- [Background] Ralston SH, Gallacher SJ, Patel U, Dryburgh FJ, Fraser WD, Cowan RA, Boyle IT. Comparison of three intravenous bisphosphonates in cancer-associated hypercalcaemia. Lancet. 1989 Nov 18;2(8673):1180-2. doi: 10.1016/s0140-6736(89)91791-1. PMID 2572902
- [Background] Cantwell BM, Harris AL. Effect of single high dose infusions of aminohydroxypropylidene diphosphonate on hypercalcaemia caused by cancer. Br Med J (Clin Res Ed). 1987 Feb 21;294(6570):467-9. doi: 10.1136/bmj.294.6570.467. PMID 3103730
- [Background] Thiebaud D, Jaeger P, Jacquet AF, Burckhardt P. Dose-response in the treatment of hypercalcemia of malignancy by a single infusion of the bisphosphonate AHPrBP. J Clin Oncol. 1988 May;6(5):762-8. doi: 10.1200/JCO.1988.6.5.762. PMID 3367184
- [Background] Guise TA. Molecular mechanisms of osteolytic bone metastases. Cancer. 2000 Jun 15;88(12 Suppl):2892-8. doi: 10.1002/1097-0142(20000615)88:12+3.0.co;2-y. PMID 10898330
- [Background] Thomas RJ, Guise TA, Yin JJ, Elliott J, Horwood NJ, Martin TJ, Gillespie MT. Breast cancer cells interact with osteoblasts to support osteoclast formation. Endocrinology. 1999 Oct;140(10):4451-8. doi: 10.1210/endo.140.10.7037. PMID 10499498
- [Background] Gucalp R, Ritch P, Wiernik PH, Sarma PR, Keller A, Richman SP, Tauer K, Neidhart J, Mallette LE, Siegel R, et al. Comparative study of pamidronate disodium and etidronate disodium in the treatment of cancer-related hypercalcemia. J Clin Oncol. 1992 Jan;10(1):134-42. doi: 10.1200/JCO.1992.10.1.134. PMID 1727915
- [Background] Nussbaum SR, Younger J, Vandepol CJ, Gagel RF, Zubler MA, Chapman R, Henderson IC, Mallette LE. Single-dose intravenous therapy with pamidronate for the treatment of hypercalcemia of malignancy: comparison of 30-, 60-, and 90-mg dosages. Am J Med. 1993 Sep;95(3):297-304. doi: 10.1016/0002-9343(93)90282-t. PMID 8368227
- [Background] Elomaa I, Blomqvist C, Grohn P, Porkka L, Kairento AL, Selander K, Lamberg-Allardt C, Holmstrom T. Long-term controlled trial with diphosphonate in patients with osteolytic bone metastases. Lancet. 1983 Jan 22;1(8317):146-9. doi: 10.1016/s0140-6736(83)92755-1. PMID 6130197
- [Background] Coleman RE, Woll PJ, Miles M, Scrivener W, Rubens RD. Treatment of bone metastases from breast cancer with (3-amino-1-hydroxypropylidene)-1,1-bisphosphonate (APD). Br J Cancer. 1988 Nov;58(5):621-5. doi: 10.1038/bjc.1988.272. PMID 3219273
- [Background] Morton AR, Cantrill JA, Pillai GV, McMahon A, Anderson DC, Howell A. Sclerosis of lytic bone metastases after disodium aminohydroxypropylidene bisphosphonate (APD) in patients with breast carcinoma. BMJ. 1988 Sep 24;297(6651):772-3. doi: 10.1136/bmj.297.6651.772. No abstract available. PMID 3142542
- [Background] Paterson AH, Powles TJ, Kanis JA, McCloskey E, Hanson J, Ashley S. Double-blind controlled trial of oral clodronate in patients with bone metastases from breast cancer. J Clin Oncol. 1993 Jan;11(1):59-65. doi: 10.1200/JCO.1993.11.1.59. PMID 8418243
- [Background] van Holten-Verzantvoort AT, Kroon HM, Bijvoet OL, Cleton FJ, Beex LV, Blijham G, Hermans J, Neijt JP, Papapoulos SE, Sleeboom HP, et al. Palliative pamidronate treatment in patients with bone metastases from breast cancer. J Clin Oncol. 1993 Mar;11(3):491-8. doi: 10.1200/JCO.1993.11.3.491. PMID 7680374
- [Background] Lahtinen R, Laakso M, Palva I, Virkkunen P, Elomaa I. Randomised, placebo-controlled multicentre trial of clodronate in multiple myeloma. Finnish Leukaemia Group. Lancet. 1992 Oct 31;340(8827):1049-52. doi: 10.1016/0140-6736(92)93075-x. PMID 1357451
- [Background] Man Z, Otero AB, Rendo P, Barazzutti L, Sanchez Avalos JC. Use of pamidronate for multiple myeloma osteolytic lesions. Lancet. 1990 Mar 17;335(8690):663. doi: 10.1016/0140-6736(90)90452-b. No abstract available. PMID 1969040
- [Background] Thiebaud D, Leyvraz S, von Fliedner V, Perey L, Cornu P, Thiebaud S, Burckhardt P. Treatment of bone metastases from breast cancer and myeloma with pamidronate. Eur J Cancer. 1991;27(1):37-41. doi: 10.1016/0277-5379(91)90056-j. PMID 1826438
- [Background] Berenson JR, Lichtenstein A, Porter L, Dimopoulos MA, Bordoni R, George S, Lipton A, Keller A, Ballester O, Kovacs MJ, Blacklock HA, Bell R, Simeone J, Reitsma DJ, Heffernan M, Seaman J, Knight RD. Efficacy of pamidronate in reducing skeletal events in patients with advanced multiple myeloma. Myeloma Aredia Study Group. N Engl J Med. 1996 Feb 22;334(8):488-93. doi: 10.1056/NEJM199602223340802. PMID 8559201
- [Background] Shipman CM, Rogers MJ, Apperley JF, Graham R, Russell G, Croucher PI. Anti-tumour activity of bisphosphonates in human myeloma cells. Leuk Lymphoma. 1998 Dec;32(1-2):129-38. doi: 10.3109/10428199809059253. PMID 10037008
- [Background] Hortobagyi GN, Theriault RL, Porter L, Blayney D, Lipton A, Sinoff C, Wheeler H, Simeone JF, Seaman J, Knight RD. Efficacy of pamidronate in reducing skeletal complications in patients with breast cancer and lytic bone metastases. Protocol 19 Aredia Breast Cancer Study Group. N Engl J Med. 1996 Dec 12;335(24):1785-91. doi: 10.1056/NEJM199612123352401. PMID 8965890
- [Background] Conte PF, Latreille J, Mauriac L, Calabresi F, Santos R, Campos D, Bonneterre J, Francini G, Ford JM. Delay in progression of bone metastases in breast cancer patients treated with intravenous pamidronate: results from a multinational randomized controlled trial. The Aredia Multinational Cooperative Group. J Clin Oncol. 1996 Sep;14(9):2552-9. doi: 10.1200/JCO.1996.14.9.2552. PMID 8823335
- [Background] Schenk R, Eggli P, Fleisch H, Rosini S. Quantitative morphometric evaluation of the inhibitory activity of new aminobisphosphonates on bone resorption in the rat. Calcif Tissue Int. 1986 Jun;38(6):342-9. doi: 10.1007/BF02555748. PMID 3089557
- [Background] Boonekamp PM, Lowik CW, van der Wee-Pals LJ, van Wijk-van Lennep ML, Bijvoet OL. Enhancement of the inhibitory action of APD on the transformation of osteoclast precursors into resorbing cells after dimethylation of the amino group. Bone Miner. 1987 Feb;2(1):29-42. PMID 3504722
- [Background] Flanagan AM, Chambers TJ. Inhibition of bone resorption by bisphosphonates: interactions between bisphosphonates, osteoclasts, and bone. Calcif Tissue Int. 1991 Dec;49(6):407-15. doi: 10.1007/BF02555852. PMID 1840176
- [Background] Reitsma PH, Teitelbaum SL, Bijvoet OL, Kahn AJ. Differential action of the bisphosphonates (3-amino-1-hydroxypropylidene)-1,1-bisphosphonate (APD) and disodium dichloromethylidene bisphosphonate (Cl2MDP) on rat macrophage-mediated bone resorption in vitro. J Clin Invest. 1982 Nov;70(5):927-33. doi: 10.1172/jci110704. PMID 7130396
- [Background] Boonekamp PM, van der Wee-Pals LJ, van Wijk-van Lennep MM, Thesing CW, Bijvoet OL. Two modes of action of bisphosphonates on osteoclastic resorption of mineralized matrix. Bone Miner. 1986 Feb;1(1):27-39. PMID 3508715
- [Background] Hughes DE, MacDonald BR, Russell RG, Gowen M. Inhibition of osteoclast-like cell formation by bisphosphonates in long-term cultures of human bone marrow. J Clin Invest. 1989 Jun;83(6):1930-5. doi: 10.1172/JCI114100. PMID 2524504
- [Background] Aparicio A, Gardner A, Tu Y, Savage A, Berenson J, Lichtenstein A. In vitro cytoreductive effects on multiple myeloma cells induced by bisphosphonates. Leukemia. 1998 Feb;12(2):220-9. doi: 10.1038/sj.leu.2400892. PMID 9519785
- [Background] Mundy GR, Raisz LG, Cooper RA, Schechter GP, Salmon SE. Evidence for the secretion of an osteoclast stimulating factor in myeloma. N Engl J Med. 1974 Nov 14;291(20):1041-6. doi: 10.1056/NEJM197411142912001. No abstract available. PMID 4413338
- [Background] O'Grady RL, Cameron DA. Osteoclasts and the resorption of bone by transplanted mammary carcinoma in rats. Br J Cancer. 1985 Jun;51(6):767-74. doi: 10.1038/bjc.1985.120. PMID 4005137
- [Background] Stewart AF, Horst R, Deftos LJ, Cadman EC, Lang R, Broadus AE. Biochemical evaluation of patients with cancer-associated hypercalcemia: evidence for humoral and nonhumoral groups. N Engl J Med. 1980 Dec 11;303(24):1377-83. doi: 10.1056/NEJM198012113032401. PMID 6253785
- [Background] Valentin-Opran A, Charhon SA, Meunier PJ, Edouard CM, Arlot ME. Quantitative histology of myeloma-induced bone changes. Br J Haematol. 1982 Dec;52(4):601-10. doi: 10.1111/j.1365-2141.1982.tb03936.x. PMID 7138789
- [Background] Taube T, Elomaa I, Blomqvist C, Beneton MN, Kanis JA. Histomorphometric evidence for osteoclast-mediated bone resorption in metastatic breast cancer. Bone. 1994 Mar-Apr;15(2):161-6. doi: 10.1016/8756-3282(94)90703-x. PMID 8086233
- [Background] Mundy GR, Ibbotson KJ, D'Souza SM. Tumor products and the hypercalcemia of malignancy. J Clin Invest. 1985 Aug;76(2):391-4. doi: 10.1172/JCI111984. No abstract available. PMID 2993358
- [Background] Garrett IR, Durie BG, Nedwin GE, Gillespie A, Bringman T, Sabatini M, Bertolini DR, Mundy GR. Production of lymphotoxin, a bone-resorbing cytokine, by cultured human myeloma cells. N Engl J Med. 1987 Aug 27;317(9):526-32. doi: 10.1056/NEJM198708273170902. PMID 3497347
- [Background] Cozzolino F, Torcia M, Aldinucci D, Rubartelli A, Miliani A, Shaw AR, Lansdorp PM, Di Guglielmo R. Production of interleukin-1 by bone marrow myeloma cells. Blood. 1989 Jul;74(1):380-7. PMID 2665838
- [Background] Russell RG, Rogers MJ. Bisphosphonates: from the laboratory to the clinic and back again. Bone. 1999 Jul;25(1):97-106. doi: 10.1016/s8756-3282(99)00116-7. PMID 10423031
- [Background] Rogers MJ, Frith JC, Luckman SP, Coxon FP, Benford HL, Monkkonen J, Auriola S, Chilton KM, Russell RG. Molecular mechanisms of action of bisphosphonates. Bone. 1999 May;24(5 Suppl):73S-79S. doi: 10.1016/s8756-3282(99)00070-8. No abstract available. PMID 10321934
- [Background] Jung A, Bornand J, Mermillod B, Edouard C, Meunier PJ. Inhibition by diphosphonates of bone resorption induced by the Walker tumor of the rat. Cancer Res. 1984 Jul;44(7):3007-11. PMID 6233002
- [Background] Radl J, Croese JW, Zurcher C, van den Enden-Vieveen MH, Brondijk RJ, Kazil M, Haaijman JJ, Reitsma PH, Bijvoet OL. Influence of treatment with APD-bisphosphonate on the bone lesions in the mouse 5T2 multiple myeloma. Cancer. 1985 Mar 1;55(5):1030-40. doi: 10.1002/1097-0142(19850301)55:53.0.co;2-y. PMID 3967188
- [Background] Nemoto R, Sato S, Nishijima Y, Miyakawa I, Koiso K, Harada M. Effects of a new bisphosphonate (AHBuBP) on osteolysis induced by human prostate cancer cells in nude mice. J Urol. 1990 Sep;144(3):770-4. doi: 10.1016/s0022-5347(17)39589-7. PMID 2117674
- [Background] Nemoto R, Satou S, Miyagawa I, Koiso K. Inhibition by a new bisphosphonate (AHBuBP) of bone resorption induced by the MBT-2 tumor of mice. Cancer. 1991 Feb 1;67(3):643-8. doi: 10.1002/1097-0142(19910201)67:33.0.co;2-w. PMID 1898709
- [Background] Sawyer N, Newstead C, Drummond A, Cunningham J. Fast (4-h) or slow (24-h) infusions of pamidronate disodium (aminohydroxypropylidene diphosphonate (APD)) as single shot treatment of hypercalcaemia. Bone Miner. 1990 May;9(2):121-8. doi: 10.1016/0169-6009(90)90078-t. PMID 2350615
- [Background] Body JJ, Magritte A, Seraj F, Sculier JP, Borkowski A. Aminohydroxypropylidene bisphosphonate (APD) treatment for tumor-associated hypercalcemia: a randomized comparison between a 3-day treatment and single 24-hour infusions. J Bone Miner Res. 1989 Dec;4(6):923-8. doi: 10.1002/jbmr.5650040617. PMID 2692407
- [Background] Body JJ, Borkowski A, Cleeren A, Bijvoet OL. Treatment of malignancy-associated hypercalcemia with intravenous aminohydroxypropylidene diphosphonate. J Clin Oncol. 1986 Aug;4(8):1177-83. doi: 10.1200/JCO.1986.4.8.1177. PMID 3016205
- [Background] Coleman RE, Rubens RD. 3(Amino-1,1-hydroxypropylidene) bisphosphonate (APD) for hypercalcaemia of breast cancer. Br J Cancer. 1987 Oct;56(4):465-9. doi: 10.1038/bjc.1987.225. PMID 3689664
- [Background] Mundy GR, Ibbotson KJ, D'Souza SM, Simpson EL, Jacobs JW, Martin TJ. The hypercalcemia of cancer. Clinical implications and pathogenic mechanisms. N Engl J Med. 1984 Jun 28;310(26):1718-27. doi: 10.1056/NEJM198406283102607. No abstract available. PMID 6328302
- [Background] Martin TJ. Humoral hypercalcemia of malignancy. Bone Miner. 1988 Apr;4(1):83-9. No abstract available. PMID 3056542
- [Background] Shinoda H, Adamek G, Felix R, Fleisch H, Schenk R, Hagan P. Structure-activity relationships of various bisphosphonates. Calcif Tissue Int. 1983;35(1):87-99. doi: 10.1007/BF02405012. PMID 6839194
- [Background] Kellihan MJ, Mangino PD. Pamidronate. Ann Pharmacother. 1992 Oct;26(10):1262-9. doi: 10.1177/106002809202601015. PMID 1421653
- [Background] Green JR, Muller K, Jaeggi KA. Preclinical pharmacology of CGP 42'446, a new, potent, heterocyclic bisphosphonate compound. J Bone Miner Res. 1994 May;9(5):745-51. doi: 10.1002/jbmr.5650090521. PMID 8053405
- [Background] Berenson JR, Vescio R, Henick K, Nishikubo C, Rettig M, Swift RA, Conde F, Von Teichert JM. A Phase I, open label, dose ranging trial of intravenous bolus zoledronic acid, a novel bisphosphonate, in cancer patients with metastatic bone disease. Cancer. 2001 Jan 1;91(1):144-54. doi: 10.1002/1097-0142(20010101)91:13.0.co;2-q. PMID 11148571
- [Background] Body JJ, Lortholary A, Romieu G, Vigneron AM, Ford J. A dose-finding study of zoledronate in hypercalcemic cancer patients. J Bone Miner Res. 1999 Sep;14(9):1557-61. doi: 10.1359/jbmr.1999.14.9.1557. PMID 10469284
- [Background] Lipton A, Small E, Saad F, Gleason D, Gordon D, Smith M, Rosen L, Kowalski MO, Reitsma D, Seaman J. The new bisphosphonate, Zometa (zoledronic acid), decreases skeletal complications in both osteolytic and osteoblastic lesions: a comparison to pamidronate. Cancer Invest. 2002;20 Suppl 2:45-54. doi: 10.1081/cnv-120014886. PMID 12442349
- [Background] Garnero P, Buchs N, Zekri J, Rizzoli R, Coleman RE, Delmas PD. Markers of bone turnover for the management of patients with bone metastases from prostate cancer. Br J Cancer. 2000 Feb;82(4):858-64. doi: 10.1054/bjoc.1999.1012. PMID 10732759
- [Background] Binkley N, Kimmel D, Bruner J, Haffa A, Davidowitz B, Meng C, Schaffer V, Green J. Zoledronate prevents the development of absolute osteopenia following ovariectomy in adult rhesus monkeys. J Bone Miner Res. 1998 Nov;13(11):1775-82. doi: 10.1359/jbmr.1998.13.11.1775. PMID 9797488
- [Background] Senaratne SG, Pirianov G, Mansi JL, Arnett TR, Colston KW. Bisphosphonates induce apoptosis in human breast cancer cell lines. Br J Cancer. 2000 Apr;82(8):1459-68. doi: 10.1054/bjoc.1999.1131. PMID 10780527
- [Background] Teronen O, Heikkila P, Konttinen YT, Laitinen M, Salo T, Hanemaaijer R, Teronen A, Maisi P, Sorsa T. MMP inhibition and downregulation by bisphosphonates. Ann N Y Acad Sci. 1999 Jun 30;878:453-65. doi: 10.1111/j.1749-6632.1999.tb07702.x. PMID 10415748
- [Background] Tassone P, Forciniti S, Galea E, Morrone G, Turco MC, Martinelli V, Tagliaferri P, Venuta S. Growth inhibition and synergistic induction of apoptosis by zoledronate and dexamethasone in human myeloma cell lines. Leukemia. 2000 May;14(5):841-4. doi: 10.1038/sj.leu.2401770. PMID 10803515
- [Background] Boissier S, Ferreras M, Peyruchaud O, Magnetto S, Ebetino FH, Colombel M, Delmas P, Delaisse JM, Clezardin P. Bisphosphonates inhibit breast and prostate carcinoma cell invasion, an early event in the formation of bone metastases. Cancer Res. 2000 Jun 1;60(11):2949-54. PMID 10850442
- [Background] Jagdev SP, Coleman RE, Shipman CM, Rostami-H A, Croucher PI. The bisphosphonate, zoledronic acid, induces apoptosis of breast cancer cells: evidence for synergy with paclitaxel. Br J Cancer. 2001 Apr 20;84(8):1126-34. doi: 10.1054/bjoc.2001.1727. PMID 11308265
- [Background] Lee MV, Fong EM, Singer FR, Guenette RS. Bisphosphonate treatment inhibits the growth of prostate cancer cells. Cancer Res. 2001 Mar 15;61(6):2602-8. PMID 11289137
- [Background] Riebeling C, Forsea AM, Raisova M, Orfanos CE, Geilen CC. The bisphosphonate pamidronate induces apoptosis in human melanoma cells in vitro. Br J Cancer. 2002 Jul 29;87(3):366-71. doi: 10.1038/sj.bjc.6600476. PMID 12177810
- [Background] Sonnemann J, Eckervogt V, Truckenbrod B, Boos J, Winkelmann W, van Valen F. The bisphosphonate pamidronate is a potent inhibitor of human osteosarcoma cell growth in vitro. Anticancer Drugs. 2001 Jun;12(5):459-65. doi: 10.1097/00001813-200106000-00007. PMID 11395574
- [Background] Mackie PS, Fisher JL, Zhou H, Choong PF. Bisphosphonates regulate cell growth and gene expression in the UMR 106-01 clonal rat osteosarcoma cell line. Br J Cancer. 2001 Apr 6;84(7):951-8. doi: 10.1054/bjoc.2000.1679. PMID 11286476
- [Background] Magnetto S, Boissier S, Delmas PD, Clezardin P. Additive antitumor activities of taxoids in combination with the bisphosphonate ibandronate against invasion and adhesion of human breast carcinoma cells to bone. Int J Cancer. 1999 Oct 8;83(2):263-9. doi: 10.1002/(sici)1097-0215(19991008)83:23.0.co;2-t. PMID 10471537
- [Background] Percival RC, Urwin GH, Harris S, Yates AJ, Williams JL, Beneton M, Kanis JA. Biochemical and histological evidence that carcinoma of the prostate is associated with increased bone resorption. Eur J Surg Oncol. 1987 Feb;13(1):41-9. PMID 3102281
- [Background] Ikeda I, Miura T, Kondo I. Pyridinium cross-links as urinary markers of bone metastases in patients with prostate cancer. Br J Urol. 1996 Jan;77(1):102-6. doi: 10.1046/j.1464-410x.1996.82817.x. PMID 8653278
- [Background] Takeuchi S, Arai K, Saitoh H, Yoshida K, Miura M. Urinary pyridinoline and deoxypyridinoline as potential markers of bone metastasis in patients with prostate cancer. J Urol. 1996 Nov;156(5):1691-5. PMID 8863572
- [Background] Clarke NW, McClure J, George NJ. Morphometric evidence for bone resorption and replacement in prostate cancer. Br J Urol. 1991 Jul;68(1):74-80. doi: 10.1111/j.1464-410x.1991.tb15260.x. PMID 1873694
- [Background] Coleman RE, Houston S, James I, Rodger A, Rubens RD, Leonard RC, Ford J. Preliminary results of the use of urinary excretion of pyridinium crosslinks for monitoring metastatic bone disease. Br J Cancer. 1992 May;65(5):766-8. doi: 10.1038/bjc.1992.161. PMID 1586605
- [Background] Vinholes J, Guo CY, Purohit OP, Eastell R, Coleman RE. Metabolic effects of pamidronate in patients with metastatic bone disease. Br J Cancer. 1996 May;73(9):1089-95. doi: 10.1038/bjc.1996.210. PMID 8624269
- [Background] Clarke NW, McClure J, George NJ. Disodium pamidronate identifies differential osteoclastic bone resorption in metastatic prostate cancer. Br J Urol. 1992 Jan;69(1):64-70. doi: 10.1111/j.1464-410x.1992.tb15461.x. PMID 1737255
- [Background] Adami S, Salvagno G, Guarrera G, Bianchi G, Dorizzi R, Rosini S, Mobilio G, Lo Cascio V. Dichloromethylene-diphosphonate in patients with prostatic carcinoma metastatic to the skeleton. J Urol. 1985 Dec;134(6):1152-4. doi: 10.1016/s0022-5347(17)47663-4. PMID 2932559
- [Background] Masud T, Slevin ML. Pamidronate to reduce bone pain in normocalcaemic patient with disseminated prostatic carcinoma. Lancet. 1989 May 6;1(8645):1021-2. doi: 10.1016/s0140-6736(89)92665-2. No abstract available. PMID 2565498
- [Background] Pelger RC, Lycklama a Nijeholt AA, Papapoulos SE. Short-term metabolic effects of pamidronate in patients with prostatic carcinoma and bone metastases. Lancet. 1989 Oct 7;2(8667):865. doi: 10.1016/s0140-6736(89)93028-6. No abstract available. PMID 2571787
- [Background] Rosen LS, Gordon D, Kaminski M, Howell A, Belch A, Mackey J, Apffelstaedt J, Hussein M, Coleman RE, Reitsma DJ, Seaman JJ, Chen BL, Ambros Y. Zoledronic acid versus pamidronate in the treatment of skeletal metastases in patients with breast cancer or osteolytic lesions of multiple myeloma: a phase III, double-blind, comparative trial. Cancer J. 2001 Sep-Oct;7(5):377-87. PMID 11693896
- [Background] Rosen LS, Gordon D, Kaminski M, Howell A, Belch A, Mackey J, Apffelstaedt J, Hussein MA, Coleman RE, Reitsma DJ, Chen BL, Seaman JJ. Long-term efficacy and safety of zoledronic acid compared with pamidronate disodium in the treatment of skeletal complications in patients with advanced multiple myeloma or breast carcinoma: a randomized, double-blind, multicenter, comparative trial. Cancer. 2003 Oct 15;98(8):1735-44. doi: 10.1002/cncr.11701. PMID 14534891
- [Background] Saad F, Gleason DM, Murray R, Tchekmedyian S, Venner P, Lacombe L, Chin JL, Vinholes JJ, Goas JA, Chen B; Zoledronic Acid Prostate Cancer Study Group. A randomized, placebo-controlled trial of zoledronic acid in patients with hormone-refractory metastatic prostate carcinoma. J Natl Cancer Inst. 2002 Oct 2;94(19):1458-68. doi: 10.1093/jnci/94.19.1458. PMID 12359855
- [Background] Saad F, Chi K, Fleshner N. The role of bisphosphonates in the management of bone metastases in prostate cancer. Can J Urol. 2004 Oct;11(5):2376-82. PMID 15576002
- [Background] Rosen LS, Gordon D, Tchekmedyian S, Yanagihara R, Hirsh V, Krzakowski M, Pawlicki M, de Souza P, Zheng M, Urbanowitz G, Reitsma D, Seaman JJ. Zoledronic acid versus placebo in the treatment of skeletal metastases in patients with lung cancer and other solid tumors: a phase III, double-blind, randomized trial--the Zoledronic Acid Lung Cancer and Other Solid Tumors Study Group. J Clin Oncol. 2003 Aug 15;21(16):3150-7. doi: 10.1200/JCO.2003.04.105. PMID 12915606
- [Background] Rosen LS, Gordon D, Tchekmedyian NS, Yanagihara R, Hirsh V, Krzakowski M, Pawlicki M, De Souza P, Zheng M, Urbanowitz G, Reitsma D, Seaman J. Long-term efficacy and safety of zoledronic acid in the treatment of skeletal metastases in patients with nonsmall cell lung carcinoma and other solid tumors: a randomized, Phase III, double-blind, placebo-controlled trial. Cancer. 2004 Jun 15;100(12):2613-21. doi: 10.1002/cncr.20308. PMID 15197804
- [Background] Major RJ, Chen BL, et al. Multiple event analysis of zoledronic acid trials in patients with cancer metastatic to bone. Proc Am Soc Clin Oncol 22:762, 2003
- [Background] Rosen LS, Gordon DH, Dugan W Jr, Major P, Eisenberg PD, Provencher L, Kaminski M, Simeone J, Seaman J, Chen BL, Coleman RE. Zoledronic acid is superior to pamidronate for the treatment of bone metastases in breast carcinoma patients with at least one osteolytic lesion. Cancer. 2004 Jan 1;100(1):36-43. doi: 10.1002/cncr.11892. PMID 14692022
- [Background] Coleman RE. Bisphosphonates: clinical experience. Oncologist. 2004;9 Suppl 4:14-27. doi: 10.1634/theoncologist.9-90004-14. PMID 15459426
- [Background] Bounameaux HM, Schifferli J, Montani JP, Jung A, Chatelanat F. Renal failure associated with intravenous diphosphonates. Lancet. 1983 Feb 26;1(8322):471. doi: 10.1016/s0140-6736(83)91465-4. No abstract available. PMID 6131186
- [Background] Kanis JA, Preston CJ, Yates AJ, Percival RC, Mundy KI, Russell RG. Effects of intravenous diphosphonates on renal function. Lancet. 1983 Jun 11;1(8337):1328. doi: 10.1016/s0140-6736(83)92434-0. No abstract available. PMID 6134112
- [Background] Harinck HI, Papapoulos SE, Blanksma HJ, Moolenaar AJ, Vermeij P, Bijvoet OL. Paget's disease of bone: early and late responses to three different modes of treatment with aminohydroxypropylidene bisphosphonate (APD). Br Med J (Clin Res Ed). 1987 Nov 21;295(6609):1301-5. doi: 10.1136/bmj.295.6609.1301. PMID 3120987
- [Background] Green JR, Seltenmeyer Y, Jaeggi KA, Widler L. Renal tolerability profile of novel, potent bisphosphonates in two short-term rat models. Pharmacol Toxicol. 1997 May;80(5):225-30. doi: 10.1111/j.1600-0773.1997.tb01964.x. PMID 9181601
- [Background] Falkmer U, Jarhult J, Wersall P, Cavallin-Stahl E. A systematic overview of radiation therapy effects in skeletal metastases. Acta Oncol. 2003;42(5-6):620-33. doi: 10.1080/02841860310014895. PMID 14596519
- [Background] Kagan AR, Rose CM, Bedwinek JM, Blitzer PH, Brascho DJ, Brown AP, Coia LR, Earle JD, Janjan NA, Lowy RO, Pieters RS Jr, Rotman M, Leibel SA. Bone metastases. American College of Radiology. ACR Appropriateness Criteria. Radiology. 2000 Jun;215 Suppl:1077-104. No abstract available. PMID 11037533
- [Background] Rose CM, Kagan AR. The final report of the expert panel for the radiation oncology bone metastasis work group of the American College of Radiology. Int J Radiat Oncol Biol Phys. 1998 Mar 15;40(5):1117-24. doi: 10.1016/s0360-3016(97)00952-8. PMID 9539567
- [Background] Chow E, Danjoux C, Wong R, Szumacher E, Franssen E, Fung K, Finkelstein J, Andersson L, Connolly R. Palliation of bone metastases: a survey of patterns of practice among Canadian radiation oncologists. Radiother Oncol. 2000 Sep;56(3):305-14. doi: 10.1016/s0167-8140(00)00238-3. PMID 10974379
- [Background] Vakaet LA, Boterberg T. Pain control by ionizing radiation of bone metastasis. Int J Dev Biol. 2004;48(5-6):599-606. doi: 10.1387/ijdb.041817lv. PMID 15349834
- [Background] Koswig S, Budach V. [Remineralization and pain relief in bone metastases after after different radiotherapy fractions (10 times 3 Gy vs. 1 time 8 Gy). A prospective study]. Strahlenther Onkol. 1999 Oct;175(10):500-8. doi: 10.1007/s000660050061. German. PMID 10554645
- [Background] Hoskin PJ, Stratford MR, Folkes LK, Regan J, Yarnold JR. Effect of local radiotherapy for bone pain on urinary markers of osteoclast activity. Lancet. 2000 Apr 22;355(9213):1428-9. doi: 10.1016/s0140-6736(00)02144-9. PMID 10791529
- [Background] Algur E, Macklis RM, Hafeli UO. Synergistic cytotoxic effects of zoledronic acid and radiation in human prostate cancer and myeloma cell lines. Int J Radiat Oncol Biol Phys. 2005 Feb 1;61(2):535-42. doi: 10.1016/j.ijrobp.2004.09.065. PMID 15667977
- [Background] Tong D, Gillick L, Hendrickson FR. The palliation of symptomatic osseous metastases: final results of the Study by the Radiation Therapy Oncology Group. Cancer. 1982 Sep 1;50(5):893-9. doi: 10.1002/1097-0142(19820901)50:53.0.co;2-y. PMID 6178497
- [Background] Blitzer PH. Reanalysis of the RTOG study of the palliation of symptomatic osseous metastasis. Cancer. 1985 Apr 1;55(7):1468-72. doi: 10.1002/1097-0142(19850401)55:73.0.co;2-m. PMID 2579716
- [Background] Price P, Hoskin PJ, Easton D, Austin D, Palmer SG, Yarnold JR. Prospective randomised trial of single and multifraction radiotherapy schedules in the treatment of painful bony metastases. Radiother Oncol. 1986 Aug;6(4):247-55. doi: 10.1016/s0167-8140(86)80191-8. PMID 3775071
- [Background] Hoskin PJ, Price P, Easton D, Regan J, Austin D, Palmer S, Yarnold JR. A prospective randomised trial of 4 Gy or 8 Gy single doses in the treatment of metastatic bone pain. Radiother Oncol. 1992 Feb;23(2):74-8. doi: 10.1016/0167-8140(92)90338-u. PMID 1372126
- [Background] Rasmusson B, Vejborg I, Jensen AB, Andersson M, Banning AM, Hoffmann T, Pfeiffer P, Nielsen HK, Sjogren P. Irradiation of bone metastases in breast cancer patients: a randomized study with 1 year follow-up. Radiother Oncol. 1995 Mar;34(3):179-84. doi: 10.1016/0167-8140(95)01520-q. PMID 7631024
- [Background] Steenland E, Leer JW, van Houwelingen H, Post WJ, van den Hout WB, Kievit J, de Haes H, Martijn H, Oei B, Vonk E, van der Steen-Banasik E, Wiggenraad RG, Hoogenhout J, Warlam-Rodenhuis C, van Tienhoven G, Wanders R, Pomp J, van Reijn M, van Mierlo I, Rutten E. The effect of a single fraction compared to multiple fractions on painful bone metastases: a global analysis of the Dutch Bone Metastasis Study. Radiother Oncol. 1999 Aug;52(2):101-9. doi: 10.1016/s0167-8140(99)00110-3. PMID 10577695
- [Background] Lardinois D, Weder W, Hany TF, Kamel EM, Korom S, Seifert B, von Schulthess GK, Steinert HC. Staging of non-small-cell lung cancer with integrated positron-emission tomography and computed tomography. N Engl J Med. 2003 Jun 19;348(25):2500-7. doi: 10.1056/NEJMoa022136. PMID 12815135
- [Background] Even-Sapir E, Metser U, Flusser G, Zuriel L, Kollender Y, Lerman H, Lievshitz G, Ron I, Mishani E. Assessment of malignant skeletal disease: initial experience with 18F-fluoride PET/CT and comparison between 18F-fluoride PET and 18F-fluoride PET/CT. J Nucl Med. 2004 Feb;45(2):272-8. PMID 14960647
- [Background] Bienert M, McCook B, Carr BI, Geller DA, Sheetz M, Tutor C, Amesur N, Avril N. 90Y microsphere treatment of unresectable liver metastases: changes in 18F-FDG uptake and tumour size on PET/CT. Eur J Nucl Med Mol Imaging. 2005 Jul;32(7):778-87. doi: 10.1007/s00259-004-1752-1. Epub 2005 Mar 17. PMID 15772860
- [Background] Ishimori T, Saga T, Nagata Y, Nakamoto Y, Higashi T, Mamede M, Mukai T, Negoro Y, Aoki T, Hiraoka M, Konishi J. 18F-FDG and 11C-methionine PET for evaluation of treatment response of lung cancer after stereotactic radiotherapy. Ann Nucl Med. 2004 Dec;18(8):669-74. doi: 10.1007/BF02985960. PMID 15682847
- [Background] Keyes JW Jr. SUV: standard uptake or silly useless value? J Nucl Med. 1995 Oct;36(10):1836-9. No abstract available. PMID 7562051
- [Background] Zasadny KR, Wahl RL. Standardized uptake values of normal tissues at PET with 2-[fluorine-18]-fluoro-2-deoxy-D-glucose: variations with body weight and a method for correction. Radiology. 1993 Dec;189(3):847-50. doi: 10.1148/radiology.189.3.8234714.
- [Background] Hiraga T, Ueda A, Tamura D, Hata K, Ikeda F, Williams PJ, Yoneda T. Effects of oral UFT combined with or without zoledronic acid on bone metastasis in the 4T1/luc mouse breast cancer. Int J Cancer. 2003 Oct 10;106(6):973-9. doi: 10.1002/ijc.11330. PMID 12918079
- [Background] Witters LM, Crispino J, Fraterrigo T, Green J, Lipton A. Effect of the combination of docetaxel, zoledronic acid, and a COX-2 inhibitor on the growth of human breast cancer cell lines. Am J Clin Oncol. 2003 Aug;26(4):S92-7. doi: 10.1097/01.COC.0000074165.90133.40. PMID 12902864
- [Background] Kouloulias V, Matsopoulos G, Kouvaris J, Dardoufas C, Bottomley A, Varela M, Uzunoglu N, Antypas C, Metafa A, Moulopoulos A, Sandilos P, Vlahos L. Radiotherapy in conjunction with intravenous infusion of 180 mg of disodium pamidronate in management of osteolytic metastases from breast cancer: clinical evaluation, biochemical markers, quality of life, and monitoring of recalcification using assessments of gray-level histogram in plain radiographs. Int J Radiat Oncol Biol Phys. 2003 Sep 1;57(1):143-57. doi: 10.1016/s0360-3016(03)00525-x. PMID 12909227
- [Background] Schirrmeister H, Guhlmann A, Kotzerke J, Santjohanser C, Kuhn T, Kreienberg R, Messer P, Nussle K, Elsner K, Glatting G, Trager H, Neumaier B, Diederichs C, Reske SN. Early detection and accurate description of extent of metastatic bone disease in breast cancer with fluoride ion and positron emission tomography. J Clin Oncol. 1999 Aug;17(8):2381-9. doi: 10.1200/JCO.1999.17.8.2381. PMID 10561300
- [Background] Peterson JJ, Kransdorf MJ, O'Connor MI. Diagnosis of occult bone metastases: positron emission tomography. Clin Orthop Relat Res. 2003 Oct;(415 Suppl):S120-8. doi: 10.1097/01.blo.0000093051.96273.7c. PMID 14600601
- [Background] Fricke E, Machtens S, Hofmann M, van den Hoff J, Bergh S, Brunkhorst T, Meyer GJ, Karstens JH, Knapp WH, Boerner AR. Positron emission tomography with 11C-acetate and 18F-FDG in prostate cancer patients. Eur J Nucl Med Mol Imaging. 2003 Apr;30(4):607-11. doi: 10.1007/s00259-002-1104-y. Epub 2003 Feb 13. PMID 12589476